CLINICAL TRIAL: NCT01235416
Title: A Phase 1b, Open-label, Dose-finding Study of AMG 706 in Combination With Gemcitabine and Erlotinib to Treat Subjects With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20050107
Record Dates: First submitted 2010-10-29; First posted 2010-11-05 (Estimated); Last update posted 2011-01-21 (Estimated); Status verified 2011-01

CONDITIONS: Histologically or Cytologically Documented Solid Tumors
MeSH Terms: interventions — motesanib diphosphate

ARMS (3):
- AMG 706 50mg (Active Comparator): 50 mg, once daily. (Cohort 1)
  Interventions: Drug: AMG 706
- AMG 706 75mg (Active Comparator): 75 mg, twice daily. (Cohort 2)
  Interventions: Drug: AMG 706
- AMG 706 125mg (Active Comparator): 125 mg, once daily. (Cohort 3)
  Interventions: Drug: AMG 706

INTERVENTIONS:
Drug: AMG 706 — In each of these 3 planned treatment cohorts, approximately 6 evaluable subjects will be treated with gemcitabine (1000-mg/m2 intravenously over 30 minutes, once weekly starting on day 1, week 1 of cycle 1) and erlotinib (100 mg orally once daily starting on day 1, week 1 of cycle 1)

SUMMARY:
This study is an open-label, dose-finding study to determine the target or maximum-tolerated dose and to characterize the safety and pharmacokinetic profile of AMG 706 administered in combination with erlotinib with or without gemcitabine in subjects with solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically documented solid tumors
* candidates for gemcitabine and erlotinib treatment (for cohorts with gemcitabine), in the opinion of the investigator
* candidates for erlotinib treatment (for cohorts without gemcitabine), in the opinion of the investigator
* Eastern Cooperative Oncology Group (ECOG) performance score of 0 to 2 (see Appendix E)
* systolic blood pressure ≤ 145 mm Hg and diastolic blood pressure ≤ 85 mm Hg (hypertension therapy is allowed)
* at least 18 years of age when written informed consent is obtained
* before any study-specific procedure is performed, the appropriate approved written informed consent must be obtained (Section 12.1).

Exclusion Criteria:

* nonsmall-cell lung cancer with squamous-cell histology
* large central tumor lesions (ie, ≥ 3 centimeters and located adjacent to or within the hilum or mediastinum)
* direct bowel wall invasion except for primary tumors of the bowel
* evidence of active bleeding or bleeding diathesis
* total gastrectomy
* hematologic malignancies
* untreated or symptomatic brain metastases
* history or evidence of interstitial lung disease
* past or current history of second neoplasm, except for curatively treated non-melanoma skin cancer, carcinoma in situ of the cervix and other primary solid cancer with no known active disease present and no curative treatment administered for the last 3 years
* documented myocardial infarction within 1 year before study day 1
* arterial thrombosis or deep vein thrombosis within 1 year before study day 1
* unstable or uncontrolled disease/condition related to or impacting cardiac function (eg, unstable angina, congestive heart failure, New York Heart Association (NYHA) > class II [Appendix F])
* major surgical procedure within 30 days before study day 1
* known positive test for human immunodeficiency virus (HIV)
* absolute neutrophil count (ANC) < 1.5 x 109 /L
* platelet count < 100 x 109 /L or > 850 x 109 /L
* hemoglobin < 9 g/dL
* serum creatinine > 2.0 mg/dL or calculated clearance < 40 mL/minute
* albumin-adjusted serum calcium < 2.0 mmol/L (8.0 mg/dL)
* urine protein quantitative value of ≥ 30 mg/dL in urinalysis or ≥ 1+ on dipstick, unless 24-hour urine protein is < 500 mg
* aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.5 x upper limit of normal (ULN) or AST or ALT > 5.0 x ULN if the subject has documented liver metastasis or primary hepatic neoplasm
* total bilirubin > 2 x ULN (> 3 x ULN for subjects with Gilbert syndrome. Subjects with UGT1A1 promoter polymorphism, i.e. Gilbert syndrome, must be confirmed by genotyping or Invader® UGT1A1 Molecular Assay)
* prothrombin time > 2.0 international normalized ratio or partial thromboplastin time > 1.5 X ULN
* currently or previously treated with bevacizumab or small molecular inhibitors of VEGF including but not limited to SU11248 (sunitinib malate), PTK787 (vatalanib), AZD 2171, AEE-788, BAY 43- 9006 (sorafenib tosylate) and AMG 706, unless approved by Amgen
* previously treated with erlotinib
* previously treated with gemcitabine (for cohorts with gemcitabine) unless approved by Amgen
* currently treated with interferon
* systemic chemotherapy within 21 days before study day 1
* radiation therapy within 14 days before study day 1
* concurrent or prior treatment with rifampin, rifabutin, rifapentin, phenytoin, carbamazepine, or phenobarbital within 14 days before study day 1
* treatment with strong CYP 3A inhibitors or inducers (such as but not limited to ketoconazole, itraconazole, clarithromycin, erythromycin or nefazodone) or immune modulators (such as but not limited to cyclosporine and tacrolimus) 7 days before study day 1
* treatment with herbal medications containing St John's Wort within 7 days before study day 1
* treatment for systemic infection within 14 days before study day 1
* treated with > 1 mg/day of warfarin within 7 days before study day 1
* any condition which in the investigator's opinion makes the subject unsuitable for study participation
* not yet completed at least 30 days since ending other investigational device/drug trial(s), or subject is receiving other investigational treatments
* pregnant (ie, positive beta-human chorionic gonadotropin test) or is breast feeding
* not using adequate contraceptive precautions
* unable to swallow oral medications
* previously enrolled into this study
* not available for follow-up assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2005-09; Primary Completion 2008-04 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
incidence of dose-limiting toxicities | Subjects will be in this study for up to 54 weeks (ie, 2 weeks screening, 48 weeks treatment and 4 weeks follow-up) or longer if subjects are deemed to have continuous clinical benefit from the combination chemotherapy and AMG 706

SECONDARY OUTCOMES:
Incidence of adverse events (including serious and treatment-related) and significant laboratory values other than those defined as dose-limiting toxicities | Subjects will be in this study for up to 54 weeks (ie, 2 weeks screening, 48 weeks treatment and 4 weeks follow-up) or longer if subjects are deemed to have continuous clinical benefit from the combination chemotherapy and AMG 706
pharmacokinetic profiles of erlotinib and AMG 706 | Subjects will be in this study for up to 54 weeks (ie, 2 weeks screening, 48 weeks treatment and 4 weeks follow-up) or longer if subjects are deemed to have continuous clinical benefit from the combination chemotherapy and AMG 706

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Derived] Kotasek D, Tebbutt N, Desai J, Welch S, Siu LL, McCoy S, Sun YN, Johnson J, Adewoye AH, Price T. Safety and pharmacokinetics of motesanib in combination with gemcitabine and erlotinib for the treatment of solid tumors: a phase 1b study. BMC Cancer. 2011 Jul 26;11:313. doi: 10.1186/1471-2407-11-313. PMID 21791058
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com